CLINICAL TRIAL: NCT06142214
Title: Pan İmmun İnflamatuar İndeks (PIV) Ile Endometriosiz Arasındaki İlişki
Brief Title: Relationship Between Pan Immune Inflammatory Index and Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Dilara SARIKAYA KURT, Specialist Doctor, Ankara Etlik City Hospital
Other Study IDs: AESH-EK1-2023-449
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Relationship Between Pan Immune Inflammatory Index and Endometriosis and Endometriosis Stages
Keywords: endometriosis; endometriosis stages; pan immune inflammatory index
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis- Case group: Patients between the ages of 18-45, who applied to the Gynecology outpatient clinic of Etlik City Hospital and were followed up in our hospital, who were suspected of endometriosis on ultrasound or MRI or CT, and who were operated and whose postoperative pathology was compatible with endometriosis will be included in the study.
- Healthy patients-Control: Patients who underwent bilateral tubal ligation in our Gynecology Clinic and who did not have any pelvic pathology will be included as the control group.

SUMMARY:
The aim of this study was to investigate whether there is a difference in terms of pan immune inflammatory index in patients with and without endometriosis and to investigate whether there is a correlation between the severity of endometriosis and this index in patients with endometriosis. To reveal the importance of the pan immune inflammatory index in predicting the severity of the disease and to contribute to the literature by examining its relationship with a new index in this sense.

DETAILED DESCRIPTION:
Endometrosis is a common estrogen-dependent chronic inflammatory disease that causes pelvic pain and infertility. Its etiology is complex and multifactorial and several theories have been proposed to explain its pathogenesis, which are not fully understood. Endometrial cells are characterized by extensive endometrial implants outside the uterus, especially in the ovaries, ligaments and peritoneal surfaces. These implants lead to inflammation resulting in scar tissue banding, also called endometrial adhesions in advanced stages (III and IV). Endometriosis affects 10-15% of reproductive women and is associated with different symptoms such as infertility, chronic pelvic pain, dyspareunia, dysmenorrhea and abnormal uterine bleeding. The American Society for Reproductive Medicine (ASRM) categorizes it into four stages according to the size of endometriotic implants in the ovaries, peritoneum and fallopian tubes and the severity of adhesion.

Stage I: This is also known as minimal endometriosis. In stage I, superficial implants and mild adhesions may grow outside the uterus. The score for minimal endometriosis is between one and five.

Stage II: This is also known as mild endometriosis. With stage II, implants may be superficial or deep with mild adhesions. In stage II, endometriosis may be widespread and deep implants may be present. Score six to 15 for mild endometriosis between Stage III: This is also known as moderate endometriosis. With stage III deep implants are available. Adhesions may also be thin and dense. As a result, endometriosis is more common than in Stage II. The score for moderate endometriosis is between 16 and 40.

Stage IV: This is also known as severe endometriosis. With stage IV, deep implants and dense adhesions are present. There may be superficial endometriosis and thin adhesions, but the disease is more widespread than in Stage III. Any score greater than 40 indicates severe endometriosis.

The pan-immune inflammatory index (neutrophil count X monocyte count X platelet count/lymphocyte count) is a scoring system of immune inflammatory cells in peripheral blood. Although this index was first studied in malignant diseases, it has been found to be associated with non-malignant diseases in subsequent studies.

In the light of the literature, we aimed to determine the relationship between pan immune inflammatory index and endometriosis and endometriosis stages.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45
* Patients with suspected endometrosis on ultrasonography or MRI or CT
* Patients with a postoperative pathologic diagnosis of endometrioma
* Patients without pelvic pathology operated for bilateral tubal ligation

Exclusion Criteria:

* Diagnosis or evidence of systemic inflammatory disease
* Having an adnexal mass other than endometriosis
* presence of infectious disease
* Mobite obesity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients between the ages of 18-45, who applied to the Gynecology outpatient clinic of Etlik City Hospital and were followed up in our hospital, who were suspected for endometriosis on ultrasound or MRI or CT, and who were operated and whose postoperative pathology was compatible with endometrioma will be included in the study. When we look at the number of operations in our Gynecology Clinic, an average of 3 endometrioma operations are performed per week. Our study period is planned as 6 months and the number of patients is planned as 100. Patients who underwent bilateral tubal ligation in our Gynecology Clinic and who do not have any pelvic pathology will be included as the control group.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of endometriosis -Pan Immune Inflammatory Index | Pre-operative
  neutrophil count x monocyte count x platelet count/lymphocyte count

SECONDARY OUTCOMES:
Stage of endometriosis -Pan Immune Inflammatory Index | Pre-operative
  neutrophil count x monocyte count x platelet count/lymphocyte count

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
patient data is not open to access due to hospital policy. however, the principal investigator can be reached via e-mail if necessary